CLINICAL TRIAL: NCT01999751
Title: SMDC CRM-MRI Prospective Case Series
Brief Title: Study to Monitor Patients With Pacemakers or ICDs Who Undergo MRI Scans
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Principal Investigator, Michael Mollerus, Physician, Essentia Health
Other Study IDs: EH12274
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Arrhythmias, Cardiac
Keywords: Magnetic Resonance Imaging; Pacemaker, Artificial; Defibrillators, Implantable
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI Scan: Patients with implantable cardioverter-defibrillator or pacemaker who undergo an MRI scan
  Interventions: Device: MRI Scan

INTERVENTIONS:
Device: MRI Scan — Clinically indicated MRI scan of patients with pacemaker or implantable cardioverter-defibrillator in situ.

SUMMARY:
This study is a prospective, non-randomized, unblinded case series of patients with permanent pacemakers and implantable cardioverter-defibrillators undergoing medically-required magnetic resonance imaging (MRI) scanning, at St. Mary's Medical Center, Essentia Health. Patients will be enrolled over a 60-month period and followed for 12 months, with data collected to evaluate the study's primary endpoint, change in pacing thresholds over time, as well as a series of secondary endpoints, including: adverse events, symptoms, need to make pacemaker programming changes, and possible artifacts created by the pacemaker systems on the MRI scans. This study will allow for carefully monitoring of the safety MRI scanning in this population and improve practice models and protocols in the future.

DETAILED DESCRIPTION:
General Approach: This study is a prospective, non-randomized, unblinded case series of patients with permanent pacemakers or implantable cardioverter-defibrillators (ICDs) undergoing medically-required MRI scanning, followed for a 12 month period. MRI scanning will be performed using accepted, standard protocols using FDA-approved equipment.

Methods and Materials: Patients will be enrolled over a 60-month period by the Principal Investigator (PI) and/or Sub-Investigator (Sub-I), at the Regional Heart Center, located at St. Mary's Medical Center, Essentia Health, Duluth, MN, during evaluations for medically-required MRI scanning. Eligible patients includes any person with a permanent pacemaker or ICD implanted for at least 6 weeks, referred for a medically-required MRI scan by a physician not participating in the trial. ICD generators must have been market released after 2001. Both pacemaker dependent and non-dependent patients are eligible. The primary endpoint is any change greater than 1 V at a pulse width of 0.5 ms in a pacemaker or ICD lead at any time within 12 months of the MRI scan.

On the day of the MRI scan, the pacemaker or ICD will be interrogated and programmed per usual practice at Essentia Health for patients undergoing an MRI scan with device in place. Three separate baseline capture threshold measurements (V) will be obtained at a fixed pulse width of 0.5 msec. Three separate baseline measurements will also be made of lead pacing impedances (Ohms) and sensed P- or R-waves (mV) using programmer default methods. Histograms will be cleared. Leads will be programmed to bipolar modality. If the patient is not device dependent, the device will be programmed to ODO/OVO/OAO mode (monitor only) if available, otherwise it will be reprogrammed to DDI or VVI mode with a lower rate of 40 bpm with pacing outputs programmed to subthreshold levels in all leads. If the participant is device dependent, the device will be programmed to an asynchronous pacing modality (DOO/VOO) with maximum pacing output. If the patient has an ICD, therapies will be disabled. The attending investigator may alter the pacing modality during the course of the scan if he or she deems it necessary to maximize patient safety or comfort. Rate responsiveness, any rate enhancements including Ventricular Rate Regulation mode, and magnet mode will be turned off.

During MRI scanning, resuscitation equipment will be available. If the participant is pacemaker dependent, the study PI or sub-I must be in the MRI suite during the scan. If the participant is not pacemaker dependent, then a pacemaker nurse will be in the MRI suite to perform pre- and post-checks, and an electrophysiologist will be available in the building for questions and troubleshooting. Patients will be asked to report all symptoms including: palpitations; pain; heat or warmth sensation; device movement; or light-headedness.

Scans will be performed using usual protocols with standard peak Specific Absorption Rate (SAR) limitations for the scan. The MRI scans will be evaluated for any artifact created by the pacemaker system. During the scan, continuous electrocardiographic and pulse oxymetry with waveform monitoring will be performed using usual protocols. Following the scan, repeat thresholds will be performed for each lead and histograms will be obtained. Three separate capture threshold measurements (V) will be obtained immediately after the patient leaves the scanner room at a fixed pulse width of 0.5 msec. Three separate measurements will also be made immediately following the scan of the lead pacing impedances (Ohms) and sensed P- or R-waves (mV) using programmer default methods. Participants who are pacemaker dependent will undergo a one-hour post-scan check using the same threshold protocol. These one-hour post scan measurements will be performed either in the pacemaker clinic if the patient is an outpatient or in the hospital if the patient is an inpatient. Any stored events detected on the device as electromagnetic interference (EMI) artifact during the scan may be retrieved and stored to diskette for later analysis. The pacemaker or ICD will be reprogrammed to original settings prior to discharge from the MRI suite unless the attending investigator deems it necessary to alter device setting to maximize patient safety or comfort. If the patient has an ICD, the capacitor will be reformed and charge time noted prior to dismissal from the MRI suite.

Patients will be followed up in the pacemaker clinic at 3 and 12 months from the MRI scan using usual clinic protocols for device follow-up. If a patient undergoes a second MRI scan, the follow-up schedule will be set based upon the most recent MRI scan.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent Pacemaker or ICD implanted for at least 6 weeks
2. Referred for medically-required MRI scan
3. Age greater than or equal to 18 years

Exclusion Criteria:

1. ICD market released before 2001 including GDT Ventak-AV, GDT MINI-II, GDT MINI-IV, GDT MINI-III, GDT Prizm, GDT Prizm-2 and MDT GEM-I series
2. Epicardial lead or subcutaneous array
3. Device has reached elective replacement indicator (ERI) or end of life (EOL)
4. Other usual contraindications to MRI scanning
5. Known or suspected lead fracture or abandoned lead
6. Pacemaker dependent patients with an ICD that cannot be programmed to asynchronous pacing (DOO/VOO)
7. Clinical factors that are deemed by the PI or Sub-I to increase the participant's risk above an acceptable clinical threshold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person followed at St. Mary's Medical Center, Duluth, MN, with a permanent pacemaker or implantable cardioverter-defibrillator implanted for at least 6 weeks, referred for a medically-required MRI scan by a physician or provider not participating in the trial. If patients elect not to participate, they may still receive an MRI and will sign the clinical consent. If they elect not to have an MRI, they will be referred back to the ordering provider to discuss other options.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-10; Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Pacing threshold increase | 12 months
  Any change greater than 1 V at a pulse width of 0.5 msec in a pacemaker or implantable cardioverter-defibrillator lead at any time within 12 months of the MRI scan

SECONDARY OUTCOMES:
Ectopy | 1 hour
  Increased cardiac ectopy at the time of the MRI scan
Pacemaker reprogramming | 12 months
  Unanticipated pacemaker or implantable cardioverter-defibrillator reprogramming because of alterations in device behavior possibly related to the MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Mollerus, MD, Principal Investigator — Essentia Health
Locations (1):
- St. Mary's Medical Center, Duluth, Minnesota, United States

REFERENCES:
- [Background] Hayes DL, Holmes DR Jr, Gray JE. Effect of 1.5 tesla nuclear magnetic resonance imaging scanner on implanted permanent pacemakers. J Am Coll Cardiol. 1987 Oct;10(4):782-6. doi: 10.1016/s0735-1097(87)80270-x. PMID 3655146
- [Background] Goldschlager N, Epstein A, Friedman P, Gang E, Krol R, Olshansky B; North American Society of Pacing and Electrophysiology (NASPE) Practice Guideline Committee. Environmental and drug effects on patients with pacemakers and implantable cardioverter/defibrillators: a practical guide to patient treatment. Arch Intern Med. 2001 Mar 12;161(5):649-55. doi: 10.1001/archinte.161.5.649. No abstract available. PMID 11231696
- [Background] Martin ET, Coman JA, Shellock FG, Pulling CC, Fair R, Jenkins K. Magnetic resonance imaging and cardiac pacemaker safety at 1.5-Tesla. J Am Coll Cardiol. 2004 Apr 7;43(7):1315-24. doi: 10.1016/j.jacc.2003.12.016. PMID 15063447
- [Background] Erlebacher JA, Cahill PT, Pannizzo F, Knowles RJ. Effect of magnetic resonance imaging on DDD pacemakers. Am J Cardiol. 1986 Feb 15;57(6):437-40. doi: 10.1016/0002-9149(86)90768-x. PMID 3946261
- [Background] Fetter J, Aram G, Holmes DR Jr, Gray JE, Hayes DL. The effects of nuclear magnetic resonance imagers on external and implantable pulse generators. Pacing Clin Electrophysiol. 1984 Jul;7(4):720-7. doi: 10.1111/j.1540-8159.1984.tb05602.x. PMID 6205375
- [Background] Sommer T, Vahlhaus C, Lauck G, von Smekal A, Reinke M, Hofer U, Block W, Traber F, Schneider C, Gieseke J, Jung W, Schild H. MR imaging and cardiac pacemakers: in-vitro evaluation and in-vivo studies in 51 patients at 0.5 T. Radiology. 2000 Jun;215(3):869-79. doi: 10.1148/radiology.215.3.r00jn08869. PMID 10831713
- [Background] Shellock FG, O'Neil M, Ivans V, Kelly D, O'Connor M, Toay L, Crues JV. Cardiac pacemakers and implantable cardioverter defibrillators are unaffected by operation of an extremity MR imaging system. AJR Am J Roentgenol. 1999 Jan;172(1):165-70. doi: 10.2214/ajr.172.1.9888762.
- [Background] Roguin A, Zviman MM, Meininger GR, Rodrigues ER, Dickfeld TM, Bluemke DA, Lardo A, Berger RD, Calkins H, Halperin HR. Modern pacemaker and implantable cardioverter/defibrillator systems can be magnetic resonance imaging safe: in vitro and in vivo assessment of safety and function at 1.5 T. Circulation. 2004 Aug 3;110(5):475-82. doi: 10.1161/01.CIR.0000137121.28722.33. Epub 2004 Jul 26. PMID 15277324
- [Background] Nazarian S, Roguin A, Zviman MM, Lardo AC, Dickfeld TL, Calkins H, Weiss RG, Berger RD, Bluemke DA, Halperin HR. Clinical utility and safety of a protocol for noncardiac and cardiac magnetic resonance imaging of patients with permanent pacemakers and implantable-cardioverter defibrillators at 1.5 tesla. Circulation. 2006 Sep 19;114(12):1277-84. doi: 10.1161/CIRCULATIONAHA.105.607655. Epub 2006 Sep 11. PMID 16966586
- [Background] Gimbel JR, Kanal E, Schwartz KM, Wilkoff BL. Outcome of magnetic resonance imaging (MRI) in selected patients with implantable cardioverter defibrillators (ICDs). Pacing Clin Electrophysiol. 2005 Apr;28(4):270-3. doi: 10.1111/j.1540-8159.2005.09520.x. PMID 15826257
- [Background] Mollerus M, Albin G, Lipinski M, Lucca J. Magnetic resonance imaging of pacemakers and implantable cardioverter-defibrillators without specific absorption rate restrictions. Europace. 2010 Jul;12(7):947-51. doi: 10.1093/europace/euq092. Epub 2010 Mar 30. PMID 20353963
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340